CLINICAL TRIAL: NCT04453709
Title: Reducing Stress, Anxiety, and Depressive Symptoms Via a Family-centered Preventative Intervention for Immigrants: A Randomized Controlled Feasibility Trial
Brief Title: Family-centered Mental Health Promotion Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Amherst (Other)
Collaborators: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Kalpana Poudel-Tandukar, Assistant Professor, University of Massachusetts, Amherst
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1837
Record Dates: First submitted 2020-06-23; First posted 2020-07-01 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-07

CONDITIONS: Stress, Psychological; Stress, Physiological; Anxiety; Depression
Keywords: Stress; Anxiety; Depression; Preventative Intervention
MeSH Terms: conditions — Stress, Psychological; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Problem Management Plus for Immigrants at family settings (Experimental): PMP-I intervention aims to develop skills in coping adaptively in a new culture, seeking help and support for mental health problems, and other life skills opportunities that can help to improve their quality of life. PMP-I intervention includes stress management through breathing exercises and yoga, problem solving, behavioral activation, and skills to strengthen social support.
  Interventions: Behavioral: Problem Management Plus for Immigrants at family settings
- Talk program with Community Support Service Pamphlet (CSS) (Active Comparator): Family receives pamphlet including list of community support service institutions that provide various health and well-being services.
  Interventions: Behavioral: Talk program with Community Support Service Pamphlet (CSS)

INTERVENTIONS:
Behavioral: Problem Management Plus for Immigrants at family settings — PMP-I is a 5-week, peer-led, culturally tailored psychoeducation, behavioral activation (90 minutes), breathing and yoga intervention (90 minutes) in a family setting. PMP-I will use a structured approach, including once a week face-to-face sessions, breathing and yoga practices.
  1. Managing Stress: Breathing and yoga practices, stress-management sessions, and behavioral activation exercises to strengthen positive coping strategies.
  2. Managing Problems: Practice exercises to identify the problems, develop solutions, and plan a strategy to carry out those solutions.
  3. Get Going, Keep Doing: Communication skill sessions and practice exercises to identify and carry out pleasant tasks.
  4. Strengthening Social Support: Social skills session and practice exercise to identify social support.
  5. Staying Well: Make a plan that helps to create supportive family environment.
  Arms: Problem Management Plus for Immigrants at family settings
Behavioral: Talk program with Community Support Service Pamphlet (CSS) — Pamphlet including list of community support service institutions
  Arms: Talk program with Community Support Service Pamphlet (CSS)

SUMMARY:
Goal: The long-term goal of the proposed research program is to test the effectiveness of a preventative behavioral intervention and to scale it up for use with broader immigrant populations to reduce stress and mental health disorders.

Intervention: This study plan to adapt the World Health Organization developed Problem Management Plus (PMP), an evidence based, multi-component, behavioral intervention including breathing, problem solving, behavioral activation, and social support for immigrants.

Hypothesis: Immigrants in the Problem Management Plus for Immigrants (PMP-I) will have significantly lower levels of stress and anxious/depressive symptoms as compared to immigrants in the talk program with Community Support Service pamphlets (CSS).

Objective: The current study aims to pilot test the feasibility and acceptability of PMP-I among Bhutanese immigrants 18 years and older living in the Massachusetts.

DETAILED DESCRIPTION:
Problem Management Plus (PMP) is a low-intensity evidence-based psychological intervention developed by World Health Organization that can be delivered by trained lay people. PMP systematically teaches four strategies: stress management through breathing exercises, problem solving, behavioral activation, and skills to strengthen social support at individual level. The current study plans to adapt PMP to develop the PMP for Immigrants (PMP-I) for a family setting to address immigrant's multiple social and emotional stressors while adjusting into the new multi-cultural environment of the United States. The rationale to adapt PMP is based on our intervention model that demands integration of social and emotional stressors; promising results of PMP; strong evidence of family and community ties in health care process; and growing consensus among community, scientists, and policymakers on the need for family-based care models that are sustainable. PMP-I is a 5-week, peer-led, culturally tailored mental health promotion program that includes psychoeducation, behavioral activation, and problem solving (90 minutes/session/weekly), and breathing exercises and yoga (90 minutes/session/weekly) in a family setting. Participating families will be randomly allocated into two groups (N=116 families (232 participants: two eligible members per family); 58 families per intervention (PMP-I) and control (CSS)) with assessments at baseline, post-intervention, and 3-month post-intervention with trained community facilitators in collaboration with church leaders.

ELIGIBILITY:
Inclusion Criteria:

* Bhutanese adult 18 years or older resettled in Massachusetts
* Have a score of 14 or below on the Patient Health Questionnaire (PHQ-9)

Exclusion Criteria:

* Have a PHQ-9 score of 15 or above
* Clinically diagnosed mental health disorders
* Taking psychiatric medications for any mental health problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Massachusetts Amherst, Amherst, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlies published results will be shared after deidentification.
Supporting Information: ICF
Time Frame: IPD will be made available after the main findings from the final research data set have been accepted for publication. No end date.
Access Criteria: Access to IPD can be requested by qualified researchers engaging in independent scientific research, and will be disseminated in accordance with University/Participating institutional and NIH policies, including entering into a Data Sharing Agreement. Inquiries for should be sent to the Principal Investigator.
URL: https://grants.nih.gov/grants/policy/data_sharing/

REFERENCES:
- [Derived] Poudel-Tandukar K, Jacelon CS, Martell CR, Poudel KC, Rai S, Ramdam R, Laws H, Meyer JS, Bertone-Johnson ER, Hollon SD. Peer-led family-centred problem management plus for immigrants (PMP-I) for mental health promotion among immigrants in USA: protocol for a pilot, randomised controlled feasibility trial. BMJ Open. 2022 May 3;12(5):e061353. doi: 10.1136/bmjopen-2022-061353. PMID 35504635

RESULTS

PARTICIPANT FLOW:
Groups:
- Problem Management Plus for Immigrants at Family Settings: PMP-I intervention aims to develop skills in coping adaptively in a new culture, seeking help and support for mental health problems, and other life skills opportunities that can help to improve their quality of life. PMP-I intervention includes stress management through breathing exercises and yoga, problem solving, behavioral activation, and skills to strengthen social support.
  Problem Management Plus for Immigrants at family settings: PMP-I is a 5-week, peer-led, culturally tailored psychoeducation, behavioral activation (90 minutes), breathing and yoga intervention (90 minutes) in a family setting. PMP-I will use a structured approach, including once a week face-to-face sessions, breathing and yoga practices.
  1. Managing Stress: Breathing and yoga practices, stress-management sessions, and behavioral activation exercises to strengthen positive coping strategies.
  2. Managing Problems: Practice exercises to identify the problems, develop solutions, and plan a strategy to carry out those solutions.
  3. Get Going, Keep Doing: Communication skill sessions and practice exercises to identify and carry out pleasant tasks.
  4. Strengthening Social Support: Social skills session and practice exercise to identify social support.
  5. Staying Well: Make a plan that helps to create supportive family environment.
Period: Overall Study
Arm/Group | Problem Management Plus for Immigrants at Family Settings | Talk Program With Community Support Service Pamphlet (CSS)
Started | 116 | 116
Completed | 116 | 116
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Problem Management Plus for Immigrants at Family Settings | Talk Program With Community Support Service Pamphlet (CSS) | Total
Number analyzed (Participants) | 116 | 116 | 232
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.60 (16.35) | 39.98 (15.46) | 41.79 (15.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 65 | 129
  Male | 52 | 51 | 103
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 116 | 116 | 232
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 116 | 116 | 232
Ever Married [Count of Participants; unit: Participants] | 104 | 94 | 198
Ever Been to School [Count of Participants; unit: Participants] | 63 | 62 | 125
Employed [Count of Participants; unit: Participants] | 59 | 58 | 117
Ever Drunk Alcohol [Count of Participants; unit: Participants] | 23 | 17 | 40
Ever Smoked [Count of Participants; unit: Participants] | 25 | 24 | 49
History of Chronic Disease [Count of Participants; unit: Participants] | 31 | 15 | 46
Duration of living in US [Mean (Standard Deviation); unit: years] | 9.45 (1.89) | 8.77 (2.26) | 9.11 (2.10)
Body weight in kg [Mean (Standard Deviation); unit: kg] | 66.93 (11.33) | 64.88 (11.80) | 65.91 (11.59)
Body height in cms [Mean (Standard Deviation); unit: cms] | 156.2 (13.34) | 157.7 (11.21) | 156.9 (12.32)
Body waist in inches [Mean (Standard Deviation); unit: inches] | 36.78 (3.88) | 35.35 (4.02) | 36.10 (4.03)
Systolic Blood Pressure [Mean (Standard Deviation); unit: millimeters of mercury] | 127.8 (11.9) | 126 (14.7) | 126.8 (13.4)
Dystolic Blood Pressure [Mean (Standard Deviation); unit: millimeters of mercury] | 84.25 (7.69) | 81.85 (7.85) | 83.05 (7.85)

OUTCOME MEASURES:

1. Primary Outcome: Cohen Perceived Stress Scale to Measure Stress
Description: The 10-item Cohen Perceived Stress Scale will be used to assess perceived stress at baseline, post-intervention, and 12-week post-intervention. The Cohen Perceived Stress Scale uses a 5-point Likert scale (ranging from 0, "never" to 4, "very often") to assess psychological stress experienced during the past four weeks, including the extent to which situations felt unpredictable, uncomfortable, and overwhelming. The total high scores indicate a worse outcome. The score range is between 0 and 40.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Problem Management Plus for Immigrants at Family Settings | Talk Program With Community Support Service Pamphlet (CSS)
Number analyzed (Participants) | 116 | 116
score on a scale | 23.28 (3.70) | 19.31 (4.87)

2. Primary Outcome: Hopkins Symptom Checklist-25 to Measure Anxiety
Description: The Hopkins Symptom Checklist-25 (HSCL-25) will be used to measure anxiety and depressive symptoms experienced over the past four weeks at baseline, post-intervention, and 12-week post-intervention. It is composed of a 10-item subscale for anxiety and a 15-item subscale for depression, with each item scored on a Likert scale from 1 (not at all) to 4 (extremely). The higher scores indicate high anxiety or depressive symptoms. The scores range for anxiety between 10 and 40 and depressive symptoms between 15 and 60.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Problem Management Plus for Immigrants at Family Settings | Talk Program With Community Support Service Pamphlet (CSS)
Number analyzed (Participants) | 116 | 116
score on a scale | 21.57 (3.25) | 15.37 (5.08)

3. Primary Outcome: Hopkins Symptom Checklist-25 to Measure Depressive Symptoms
Description: as for outcome 2
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Problem Management Plus for Immigrants at Family Settings | Talk Program With Community Support Service Pamphlet (CSS)
Number analyzed (Participants) | 116 | 116
score on a scale | 32.11 (4.89) | 22.56 (6.24)

4. Secondary Outcome: Hair Cortisol Concentrations (pg/mg)
Description: Cortisol hair test (average hormone levels over the past 3 months) will be used as a biomarker to measure physiological stress. Higher hair cortisol concentrations indicate a higher level of biological stress in the body. The range of values is between 0.799 and 2554.68 pg/mg.
Time Frame: Baseline
Population: Intervention Group: Only 84 participants provided hair samples out of 116 total participants.
  Control Group: Only 71 participants provided hair samples out of 116 total participants.
Measure: Mean (Standard Deviation); unit: pg/mg
Arm/Group | Problem Management Plus for Immigrants at Family Settings | Talk Program With Community Support Service Pamphlet (CSS)
Number analyzed (Participants) | 84 | 71
pg/mg | 349.37 (2627.98) | 78.35 (324.36)

ADVERSE EVENTS:
Time Frame: 41/2 months
Arm/Group | Problem Management Plus for Immigrants at Family Settings | Talk Program With Community Support Service Pamphlet (CSS)
All-Cause Mortality (participants affected / at risk) | 0/116 | 0/116
Serious Adverse Events (participants affected / at risk) | 0/116 | 0/116
Other Adverse Events (participants affected / at risk) | 0/116 | 0/116

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/09/NCT04453709/Prot_SAP_000.pdf